CLINICAL TRIAL: NCT06508983
Title: A Phase 3 Randomized, Placebo-controlled, Double-blind, Multicenter Study Comparing SG301 in Combination With Pomalidomide and Dexamethasone Versus Placebo in Combination With Pomalidomide and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Clinical Study Comparing SG301 Plus Pomalidomide and Dexamethasone to Placebo Plus Pomalidomide and Dexamethasone in Relapsed or Refractory Multiple Myeloma Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Sumgen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSG-301-301
Record Dates: First submitted 2024-07-05; First posted 2024-07-19 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: This Study consists of Stage 1 and Stage 2.
  Stage 1 ：Single group. Subjects will receive SG301 Injection in combination with pomalidomide and dexamethasone.
  Stage 2：Parallel. Subjects will be randomized to receive SG301 Injection in combination with pomalidomide and dexamethasone or placebo in combination with pomalidomide and dexamethasone.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stage 1#Open-label Stage 2#Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SG301 Injection in combination with pomalidomide and dexamethasone (Experimental): Participants will receive SG301 Injection in combination with pomalidomide and dexamethasone. Treatment cycles have a duration of 28 days. Participants will continue to receive study treatment until confirmed disease progression, unacceptable toxicity, or any other treatment discontinuation criteria are met.
  Interventions: Drug: SG301 Injection; Drug: pomalidomide; Drug: dexamethasone
- Placebo in combination with pomalidomide and dexamethasone (Placebo Comparator): Participants in Stage 2 who randomized to this arm will receive placebo in combination with pomalidomide and dexamethasone. Treatment cycles have a duration of 28 days. Participants will continue to receive study treatment until confirmed disease progression, unacceptable toxicity, or any other treatment discontinuation criteria are met.
  Interventions: Drug: SG301 placebo; Drug: pomalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: SG301 Injection — Dosage form: solution for infusion Route of administration: intravenous Frequency: weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) thereafter.
  Arms: SG301 Injection in combination with pomalidomide and dexamethasone
Drug: SG301 placebo — Dosage form: solution for infusion Route of administration: intravenous Frequency: weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) thereafter.
  Arms: Placebo in combination with pomalidomide and dexamethasone
Drug: pomalidomide — Dosage form: capsule Route of administration: oral Dosage: 4 mg Frequency: once daily on Days 1 through 21 of each 28-day cycle.
Drug: dexamethasone — Dosage form: tablets or solution for infusion Route of administration: oral or intravenous Dosage: 40 mg (participants with BMI < 18.5 kg/m2 received 20 mg dexamethasone) Frequency: once daily on Day 1, 8, 15, 22 of each 28-day treatment cycle.

SUMMARY:
The purpose of this study is to evaluate the effects of the addition of SG301 injection to pomalidomide and dexamethasone in subjects with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, multicenter phase III clinical study to compare SG301 injection in combination with pomalidomide and dexamethasone versus placebo in combination with pomalidomide and dexamethasone in patients with relapsed or refractory multiple myeloma who have received at least 1 prior treatment regimen with both lenalidomide and a proteasome inhibitor and have demonstrated disease progression.

This study consists of two stages. Stage 1 is the dose exploration stage to confirm the recommended stage 2 dose of SG301 injection in combination with pomalidomide and dexamethasone in patients with relapsed/refractory multiple myeloma. Stage 2 is the randomized controlled stage of SG301 injection in combination with pomalidomide and dexamethasone versus placebo in combination with pomalidomide and dexamethasone in patients with relapsed/refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the informed consent form (ICF).
2. Males and females aged 18-75 years (inclusive)
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1 or 2
4. Expected survival time of ≥3 months.
5. Subjects had a documented diagnosis of multiple myeloma with evidence of measurable disease.
6. Subjects had received at least 1 prior lines of anti-myeloma therapy, which must include lenalidomide and a proteasome inhibitor (bortezomib, carfilzomib or ixazomib) given alone or in combination.
7. Subjects must have documented evidence of PD on or after the last regimen.
8. Adequate function of vital organs
9. Women of childbearing potential (WOCBP) must agree to follow instructions for methods of contraception for 4 weeks before the start of study treatment, for the duration of study treatment, and for 6 months after cessation of SG301 or 4 weeks after cessation of pomalidomide, whichever is longer. WOCBP must have 2 negative serum or urine pregnancy tests, one 10-14 days prior to start of study treatment and one 24 hours prior to the start of study treatment.

Exclusion Criteria:

1. Primary refractory multiple myeloma defined as participants who had never achieved at least a minimal response (MR) with any treatment during the disease course.
2. Bone independent extramedullary disease at screening.
3. Subjects who are primary refractory to a prior CD38 monoclonal antibody therapy.
4. Previous exposure to pomalidomide.
5. Subject has received chemotherapy or small molecule antitumor therapy within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is shorter, before the first dose of study treatment;
6. Subject has received tumor biotherapy within 4 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is shorter, before the first dose of study treatment;
7. Subject has received investigational agents within 4 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is shorter (but not less than 14 days), before the first dose of study treatment;
8. Active hepatitis B, or C.
9. Known HIV infection.
10. Known active tuberculosis or positive treponema pallidum antibodies.
11. Subjects with clinical significant organ dysfunction that does not meet the study needs.
12. Previous allogenic stem cell transplant or autologous stem cell transplantation (ASCT) before the first dose of study treatment.
13. Known allergy to any component of the investigational medicinal product.
14. Any concurrent medical or psychiatric condition or disease (eg, active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with the study procedures or results or that, in the opinion of the investigator, would constitute a hazard for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events （stage 1） | From date of first dose of study intervention through approximately 30 days after last study intervention administration, assessed up to approximately 4 years.
  AEs, DLTs, laboratory abnormality, Vital signs or ECG abnormalities, ECOG scores, abnormal physical examination
Recommended stage 2 dose of SG301 (Stage 1) | Up to approximately 6 months.
  Recommended stage 2 dose of SG301 will be determined based on the DLTs and safety data
Progression Free Survival (Stage 2) | From baseline through the end of study. Assessed every 4 weeks after randomization until C19D1, and every 8 weeks thereafter until disease progression (IMWG criteria) or death whichever occurs first, assessed up to approximately 4 years.
  Comparison of Progression Free Survival between treatment arms (SG301/Pomalidomide/Dexamethasone vs Placebo/Pomalidomide/Dexamethasone).

SECONDARY OUTCOMES:
Pharmacokinetics (PK): AUC | From date of first dose of study intervention through approximately 30 days after last study intervention administration, assessed up to approximately 4 years.
  The area under the curve (AUC) of serum concentration of the drug after the administration.
Pharmacokinetics (PK): Cmax | From date of first dose of study intervention through approximately 30 days after last study intervention administration, assessed up to approximately 4 years.
  Cmax to maximum drug concentration.
Pharmacokinetics (PK):limination half-life (T1/2) | From date of first dose of study intervention through approximately 30 days after last study intervention administration, assessed up to approximately 4 years.
  Limination half-life (T1/2) of the drug after administration.
Immunogenicity endpoints | From date of first dose of study intervention through approximately 30 days after last study intervention administration, assessed up to approximately 4 years.
  Anti-SG301 antibody, neutralizing antibody (to be detected only in case of the presence of anti-SG301 antibody.
Overall Response Rate | From baseline through the end of study. It is measured from the start of treatment until disease progression, death, initiation of further anti-myeloma treatment, or cut-off date, whichever occurs first, assessed up to approximately 4 years.
  ORR (IMWG criteria): percentage of participants with stringent complete response(sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) as best overall response
Percentage of Participants With Very Good Partial Response (VGPR) or Better (≥VGPR Rate) | From baseline through the end of study. It is measured from the start of treatment until disease progression, death, initiation of further anti-myeloma treatment, or cut-off date, whichever occurs first, assessed up to approximately 4 years.
  ≥VGPR Rate (IMWG criteria): percentage of participants with stringent complete response(sCR), complete response (CR), and very good partial response (VGPR) as best overall response.
Duration of Response | From baseline through the end of study. It is measured from the time that the criteria for objective response are first met until the date of a progression event, assessed up to approximately 4 years.
  Duration of response will be restricted to subjects who achieve a best objective response of PR or better.
Overall Survival | From baseline through the end of study, assessed up to approximately 4 years.
  Overall survival is defined as the time, in months, from randomization to the date of death from any cause.
Percentage of Participants With Minimal Residual Disease (MRD) | From baseline through the end of study. It is measured from the time that the criteria for CR are first met until the date of a progression event, assessed up to approximately 4 years.
  MRD was assessed by next-generation sequencing in bone marrow samples from participants who achieved CR or sCR, to determine the depth of response at the molecular level.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Beijing Chaoyang Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital Of Soochow University, Suzhou, Jiangsu
  - Shanxi Provincial Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital Of Xi an Jiaotong University (Xibei Hospital), Xi’an, Shanxi
  - Tianjin Cancer University Airport Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang